CLINICAL TRIAL: NCT04633421
Title: The Impact of High Versus Standard Enteral Protein Provision on Functional Recovery Following Intensive Care Admission: a Randomized Controlled, Multicenter, Parallel Group Trial in Mechanically Ventilated, Critically Ill Patients
Brief Title: PRotEin Provision in Critical IllneSs
Acronym: PRECISe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other); Zuyderland Medisch Centrum (Other); Gelderse Vallei Hospital (Other); Medisch Spectrum Twente (Other); Centre Hospitalier Universitaire de Liege (Other); Centre Hospitalier Régional de la Citadelle (Other); Universitair Ziekenhuis Brussel (Other); General Hospital Groeninge (Other); Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL73247.068.20; 80-85200-98-18574 (Other Grant/Funding Number: KCE-ZonMW (BeNeFIT))
Record Dates: First submitted 2020-10-23; First posted 2020-11-18 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Critical Illness; Intensive Care Unit Acquired Weakness
Keywords: Enteral Nutrition; Dietary Proteins; Respiratory failure; Catabolism
MeSH Terms: conditions — Critical Illness; Respiratory Insufficiency | interventions — Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study feeds will be blinded. Dosing of intervention will be volume based, with the same volume targets for both groups. Differences in composition of study feeds will result in differences in protein intake at similar volume administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRECISe protocol EN (8g protein/100kcal) (Experimental): Enteral (EN) feed with 8 grams protein per 100 kcal (2.0 g/kg/day protein when on target). The caloric goal is 25 kcal/kg/day to be reached on day 4 of ICU admission.
  Interventions: Dietary Supplement: PRECISe protocol EN 8g protein/100kcal
- PRECISe protocol EN (5g protein/100kcal) (Active Comparator): Enteral (EN) feed with 5 grams protein per 100 kcal (1.3 g/kg/day protein when on target). The caloric goal is 25 kcal/kg/day to be reached on day 4 of ICU admission.
  Interventions: Dietary Supplement: PRECISe protocol EN 5g protein/100kcal

INTERVENTIONS:
Dietary Supplement: PRECISe protocol EN 8g protein/100kcal — Enteral feed containing 8g protein/100kcal
  Arms: PRECISe protocol EN (8g protein/100kcal)
Dietary Supplement: PRECISe protocol EN 5g protein/100kcal — Enteral feed containing 5g protein/100kcal
  Arms: PRECISe protocol EN (5g protein/100kcal)

SUMMARY:
Rapid skeletal muscle wasting during critical illness had a detrimental impact on both short and long term outcomes following ICU admission. Increased dietary protein delivery might attenuate skeletal muscle wasting and its subsequent effects on post-ICU function.

The investigators will conduct a 935 patient, randomised controlled, quadruple blinded parallel group trial to determine whether enteral nutrition with increased protein content in mechanically ventilated, critically ill patients is able to improve functional recovery.

DETAILED DESCRIPTION:
ICU-acquired weakness (ICU-AW) is frequent among ICU survivors and negatively affects both short and long term outcomes. ICU-AW is the consequence of the body's reserves being depleted during critical illness and results in severe skeletal muscle wasting during the first week of ICU admission.Therefore, measures aimed at preserving muscle mass during critical illness and improving recovery after ICU discharge are urgently needed.

Retrospective observational cohort studies suggest that the administration of high protein nutrition is associated with improved survival and outcome. Current ICU guidelines recommend dietary protein delivery at 1.3 g/kg/day (ESPEN), or even up to 2.0 g/kg/day (ASPEN). However, strong prospective clinical evidence on the effectiveness and safety of high enteral protein delivery is lacking and urgently awaited. Therefore, the aim of the present study is to investigate the effect of high versus standard protein provision on the functional recovery of critically ill patients.

The focus on functional, patient-centered outcomes rather than traditional clinical endpoints like mortality is an important aspect and strength of the study. Previous nutritional intervention studies focusing primarily on improving mortality have repeatedly shown no effect. Therefore, it is nowadays increasingly recognized to move primary ICU trial endpoints away from classical outcomes, such as survival or length of stay, towards more functional outcomes, in line with the underlying pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or above) patient admitted to the ICU
* Unplanned ICU admission
* Invasive mechanical ventilation initiated <24 hours of ICU admission
* Expected ICU stay on ventilator support of 3 days or more

Exclusion Criteria:

* Contraindication for enteral nutrition
* Moribund or expected withholding of treatment
* Kidney failure AND 'no-dialysis'-code on admission
* Hepatic encephalopathy.(West Haven grade 3 or 4)
* Body-mass index < 18 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 935 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life (HRQL) | Day 0, Day 30, 90 and 180 after index ICU admission.
  Overall difference in EQ-5D single summary index between intervention and control group over the three time-points combined, corrected for baseline. A higher summary index indicates better Health related Quality of Life.

SECONDARY OUTCOMES:
Overall survival | Day 30, 90 and 180 after ICU admission
  Overall survival
Health-related Quality of Life - SF-36 | Day 30, 90 and 180 after ICU admission
  Short Form 36 (SF-36), ranging from 0 to 100. A higher score indicates a better Health-related Quality of Life.
Mental health status - anxiety/depression | Day 30, 90 and 180 after ICU admission
  Hospital Anxiety and Depression Scale (HADS), ranging from 0 to 42. Questions 1, 3, 5, 7, 9, 11 and 13 measure symptoms of anxiety (range: 0-21). Questions 2, 4, 6, 8, 10, 12 and 14 measure symptoms of depression (range: 0-21). Higher scores indicate worse symptoms of anxiety and depression.
Pain intensity | Day 0, Day 30, 90 and 180 after index ICU admission
  EQ-5D pain question, ranging from 1 to 5, corrected for baseline. A higher score indicates a more severe perception of pain.
Self-reported health | Day 0, Day 30, 90 and 180 after index ICU admission
  EQ-5D Visual Analogue Scale (EQ-VAS), ranging from 0 to 100. A higher score indicates a better self-reported health.
Mental health status - post-traumatic stress | Day 30, 90 and 180 after ICU admission.
  Impact of Event Scale Revised (IES-R), ranging from 0 to 88. A higher score indicates worse symptoms of Post-Traumatic Stress Disorder.
Physical function - 6-minute walk test | Day 30, 90 and 180 after ICU admission
  6-minute walk test. Data collected during 6-minute walk test are pre- and post-test saturation and pulse and total distance walked with or without the use of any aids.
Muscle and nerve function - MRC-sum score | Day 30, 90 and 180 after ICU admission
  Medical Research Council (MRC-)sum score, ranging from 0 to 60. A higher score indicates better muscle and nerve function.
Muscle and nerve function - handgrip strength | Day 30, 90 and 180 after ICU admission.
  Handgrip strength, assessed via a hand dynamometer and measured in kilograms (kg).

OTHER OUTCOMES:
Duration of mechanical ventilation | During index ICU stay, up to 90 days.
  Number of days on invasive mechanical ventilation.
Duration of index ICU stay | During index ICU stay, up to 90 days.
  Number of days in ICU.
Duration of index hospital stay | From date of randomization until the date of index hospital discharge, assessed up to 6 months.
  Number of days in hospital.
Hospital mortality | From index ICU admission until index hospital discharge, assessed up to 6 months.
  Hospital mortality
30-day mortality | From index ICU admission until day 30.
  Mortality at 30 days after ICU admission.
60-day mortality | From index ICU admission until day 60.
  Mortality at 60 days after ICU admission.
90-day mortality | From index ICU admission until day 90.
  Mortality at 90 days after ICU admission.
Time-to-discharge-alive | From index ICU admission until index hospital discharge, assessed up to 6 months.
  Days until live hospital discharge
Days alive and at home at day 90 | From index ICU admission until day 90.
  Number of days alive and at home at day 90 after ICU admission.
Nutritional adequacy | From index ICU admission until index ICU discharge, assessed up to 6 months.
  Ratio between total amount of calories and grams of protein actually received by patients and prescribed during treatment period.
Administration of prokinetics | During index ICU stay, up to 90 days.
  Number of patients who received a prokinetic and number of days on it.
Incidence of gastrointestinal intolerance/symptoms | During index ICU stay, up to 90 days.
  Number of patients that experienced gastrointestinal intolerance or symptoms at any time during index ICU stay, i.e. vomiting, ischemia, diarrhea, abdominal distention, gastric paresis, bleeding/ulcer.
Incidence of ICU-readmission | From date of randomization until the date of index hospital discharge, assessed up to 6 months.
  Number of patients readmitted to the ICU during index hospital stay and number of readmissions per patient.
Incidence of ICU-acquired infections | During index ICU stay, up to 90 days.
  Number of patients who contracted an ICU-acquired infection.
Incidence of acute kidney injury | During index ICU stay, up to 90 days.
  Number of patients with Acute Kidney Injury (AKI), defined as a serum creatinine level higher than 2 times baseline level.
Incidence and duration of renal replacement therapy | During index ICU stay, up to 90 days.
  Number of patients who received renal replacement therapy and days on it.
Incidence of hepatic dysfunction | During index ICU stay, up to 90 days.
  Number of patients with hepatic dysfunction, defined as a total bilirubin level > 3mg/dL.
Maximum and mean SOFA score | During index ICU stay, up to 90 days.
  Sequential Organ Failure Assessment score (SOFA), ranging from 0 to 24. A higher score indicates more severe multi-organ failure.
Difference in mobilization treatment | During index ICU stay, up to 90 days.
  Number of days and degree of daily mobilization (passive/active, in-bed cycling etc).
Difference in frailty | Day 0, Day 30, 90 and 180 after index ICU admission.
  Rockwood Clinical Frailty Scale, ranging from 1 to 9, corrected for baseline. A higher score indicates a more severe degree of frailty.
Domain data EQ-5D | Day 30, 90 and 180 after ICU admission.
  Scores of subdomains of EQ-5D, ranging from 1 to 5. A higher score indicates a higher severity level on that subdomain.
Destination of hospital discharge | Follow-up until 180 days after index ICU admission.
  Destination of hospital discharge (home, rehabilitation center, care facility etc).
Length of stay at rehabilitation facility | Follow-up until 180 days after index ICU admission.
  Number of days at rehabilitation center.
Time to return to work | Follow-up until 180 days after index ICU admission.
  Number of days between ICU admission and return to work.
Health economic analysis | From index ICU admission until 180 days.
  Total health care costs.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel CG van de Poll, MD, PhD, Principal Investigator — Maastricht UMC
Locations (10):
- Belgium (5):
  - UZ Brussel, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - AZ Groeninge, Kortrijk
  - CHR de la Citadelle, Liège
  - CHU Liège, Liège
- Netherlands (5):
  - Catharina Ziekenhuis Eindhoven, Eindhoven, North Brabant
  - Gelderse Vallei Ede, Ede
  - Medisch Spectrum Twente, Enschede
  - Zuyderland Medisch Centrum, Heerlen
  - Maastricht Universtair Medisch Centrum, Maastricht

REFERENCES:
- [Background] Needham DM, Sepulveda KA, Dinglas VD, Chessare CM, Friedman LA, Bingham CO 3rd, Turnbull AE. Core Outcome Measures for Clinical Research in Acute Respiratory Failure Survivors. An International Modified Delphi Consensus Study. Am J Respir Crit Care Med. 2017 Nov 1;196(9):1122-1130. doi: 10.1164/rccm.201702-0372OC. PMID 28537429
- [Derived] Schouteden E, Heuts S, Bels JL, Thiesen S, van Gassel RJ, Lee ZY, Stoppe C, Beishuizen A, De Bie Dekker A, Fraipont V, Lamote S, Ledoux D, Scheeren C, De Waele E, van Zanten A, van Kuijk SM, van de Poll MC, Mesotten D, Gabrio A; PRECISe study team. The impact of high versus standard enteral protein provision on functional recovery following intensive care admission: A pre-planned Bayesian analysis of the PRECISe trial. Clin Nutr. 2025 May;48:153-160. doi: 10.1016/j.clnu.2025.03.022. Epub 2025 Apr 1. PMID 40215884
- [Derived] Bels JLM, Thiessen S, van Gassel RJJ, Beishuizen A, De Bie Dekker A, Fraipont V, Lamote S, Ledoux D, Scheeren C, De Waele E, van Zanten ARH, Bormans-Russell L, van Bussel BCT, Dictus MMJ, Fivez T, Harks I, van der Horst ICC, Jonckheer J, Marechal H, Massion PB, Meex I, Paulus MC, Rinket M, van Santen S, Tartaglia K, Deane AM, Demuydt F, Puthucheary Z, Vloet LCM, Weijs PJM, van Kuijk SMJ, van de Poll MCG, Mesotten D; PRECISe study team. Effect of high versus standard protein provision on functional recovery in people with critical illness (PRECISe): an investigator-initiated, double-blinded, multicentre, parallel-group, randomised controlled trial in Belgium and the Netherlands. Lancet. 2024 Aug 17;404(10453):659-669. doi: 10.1016/S0140-6736(24)01304-7. PMID 39153816
- [Derived] van Gassel RJJ, Bels JLM, Tartaglia K, van Bussel BCT, van Kuijk SMJ, Deane AM, Puthucheary Z, Weijs PJM, Vloet L, Beishuizen B, De Bie Dekker A, Fraipont V, Lamote S, Ledoux D, Scheeren C, De Waele E, van Zanten ARH, Mesotten D, van de Poll MCG. The impact of high versus standard enteral protein provision on functional recovery following intensive care admission (PRECISE trial): study protocol for a randomized controlled, quadruple blinded, multicenter, parallel group trial in mechanically ventilated patients. Trials. 2023 Jun 19;24(1):416. doi: 10.1186/s13063-023-07380-3. PMID 37337234

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT04633421/SAP_000.pdf